CLINICAL TRIAL: NCT02838316
Title: Muscle Cell Mediated Therapy for Tongue Dysphagia: An Investigation of Cook MyoSite Autologous Muscle Derived Cells
Brief Title: Autologous Muscle Derived Cells for Gastro-Intestinal Repair (AMDC-GIR) for Tongue Dysphagia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peter Belafsky, MD (Other)
Collaborators: Cook MyoSite (Industry)
Responsible Party: Sponsor-Investigator, Peter Belafsky, MD, Professor and Director of Voice and Swallowing Center,UC Davis Health System-Department of Otolaryngology, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 801019; 801019-1 (Other: UC Davis)
Record Dates: First submitted 2016-07-12; First posted 2016-07-20 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Oropharyngeal Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Phase I open label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 150 x 106 dosage (Experimental): 10 subjects will be receiving a dosage of 150 x 106 AMDC-GIR
  Interventions: Drug: Autologous Muscle Derived Cells for Gastro-Intestinal Repair (AMDC-GIR)
- 300 x 106 dosage (Experimental): 10 subjects will be receiving a dosage of 300 x 106 AMDC-GIR
  Interventions: Drug: Autologous Muscle Derived Cells for Gastro-Intestinal Repair (AMDC-GIR)

INTERVENTIONS:
Drug: Autologous Muscle Derived Cells for Gastro-Intestinal Repair (AMDC-GIR) — Autologous muscle derived stem cells

SUMMARY:
The primary objective of this study is to evaluate the safety of Autologous Muscle Derived Cells for Gastro-Intestinal Repair (AMDC-GIR) during the 12 months following treatment of tongue dysphagia in male and female patients who have undergone surgery and/or chemo- and/or radiotherapy for squamous cell cancer of the oropharynx.

DETAILED DESCRIPTION:
This preliminary, prospective, dose escalating clinical study will evaluate the safety and potential efficacy of Autologous Muscle Derived Cells for Gastro-Intestinal Repair (AMDC-GIR) for the treatment of tongue dysphagia (TD) that develops following treatment for head and neck cancer.

Surgery, chemo- and radiotherapy can induce significant TD resulting in long-term TD. Therefore, augmenting tongue muscle function may be beneficial to patients. Autologous muscle cell therapy, which involves isolation of cells from skeletal muscle biopsies, ex vivo expansion, and subsequent injection into the tongue, may serve as a potential durable therapy. In animal studies, muscle derived cells have successfully integrated within tissue to improve tongue strength and function. Intramuscular injection of AMDC-GIR is expected to produce localized tissue changes near the injection site and is not expected to produce a systemic effect.

Patients will receive a single treatment intramuscular injection of 1 of 2 doses of AMDC-GIR. Patients will have quantitative and qualitative measures of dysphagia assessed before treatment and at various times after treatment.

The study will treat up to 20 patients at 1 clinical site. Enrollment is expected to be completed within 2 years of initiating the study. Patients will be followed for 24 months post-treatment. The first 3 patients at each dose must reach 1-month follow-up before subsequent patients can be treated.

Male and female patients at least 18 years of age who have undergone surgery and/or chemo- and or radiotherapy for primary treatment of oropharyngeal squamous cell cancer and who present with symptoms and findings of TD will be eligible for participation. Eligible patients will have muscle tissue harvested using a needle biopsy technique during an outpatient procedure. The harvested muscle tissue will be transported to the manufacturer for cell processing. The muscle derived cells (MDC) will be isolated and expanded in culture over several weeks.

After reaching the desired concentration, the isolated and expanded AMDC-GIR will be frozen and shipped back to the investigating physician. The physician will thaw the AMDC-GIR and dilute the sample with an approximately equal volume of physiological saline. Under direct vision, the resulting suspension will be injected into the patient's tongue in a brief outpatient procedure.

Patients will be assessed for improvement in TD symptoms at 3 months, 6 months, 12 months and 24 months following treatment. Adverse events will be assessed at those visits, as well as during follow-up calls at 1-2 days, 1 week, 15 months, 18 months and 21 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, at least 18 years old, with primary symptoms of TD following surgery and/or chemo- and/or radiotherapy for treatment of squamous cell carcinoma for oropharyngeal cancer. Treatment must be completed at least 24 months prior to enrollment, with TD and disease-free status confirmed by medical history and clinical symptoms, including a focused head and neck examination evaluation, swallowing fluoroscopy, and high resolution pharyngeal manometry.
2. TD severity should be moderate as defined by a Functional Oral Intake Scale (FOIS, provided in Appendix C). Individuals must have a FOIS of 3 or better.
3. Patient has failed to achieve acceptable resolution of symptoms following conservative therapies.

Exclusion Criteria:

Patient History-based Criteria:

1. Simultaneously participating in another investigational drug or device study or has completed the follow-up phase for the primary endpoint of any previous study less than 30 days prior to the first evaluation in this study.
2. Previously treated with an investigational device, drug, or procedure for TD within 6 months prior to signing consent.
3. Has ever been treated with a cell therapy for TD.
4. Symptoms of aspiration pneumonia prior to enrollment.
5. TD of neurogenic etiology or uncorrected congenital abnormality leading to TD.
6. Neuromuscular disorder (e.g., Parkinson's disease, muscular dystrophy, multiple sclerosis) that could lead to TD.
7. Moderate or severe fibrosis at likely injection site.
8. Morbidly obese (BMI ≥ 35).
9. Uncontrolled diabetes.
10. Compromised immune system due to disease state, chronic corticosteroid use, or other immunosuppressive therapy.
11. Medical condition or disorder that may limit life expectancy or that may cause clinical investigation plan (CIP) deviations (e.g., unable to perform self-evaluations or accurately report medical history, symptoms, or data).
12. History of bleeding diathesis or uncorrectable coagulopathy.
13. Known allergy or hypersensitivity to bovine proteins or allergens, gentamicin sulfate, or ampicillin that medically warrants exclusion as determined by the physician.
14. Any non-skin cancer that has necessitated treatment within the past 24 months.

Patient's Current Status-based Criteria:

1. Evidence or known high risk of recurrent or persistent cancer as determined by the physician during screening.
2. Tests positive for Hepatitis B (required tests: Hepatitis B Surface Antigen [HBsAg] and Anti-Hepatitis B Core Antibody [Anti-HBc]), Hepatitis C (required test: Hepatitis C Antibody [Anti-HCV]), HIV (required tests: HIV Type 1 and 2 Antibodies [Anti-HIV-1, 2]), and/or Syphilis.

   a. Tests performed by certified/authorized testing laboratory using licensed/approved tests and performed on blood samples collected within 30 days prior to muscle tissue procurement.
3. Cannot, or is not willing to, maintain the current treatment regimen for existing conservative therapy (e.g., swallowing therapy).
4. Requires prophylactic antibiotics for chronic infections, or has required 2 or more courses of antibiotics for infections in the 2 months prior to signing consent.
5. Any condition, including current infection, which could lead to significant postoperative complications.
6. Refuses to provide written informed consent.
7. Not available for, or willing to comply, with the baseline and follow-up evaluations as required by the CIP.
8. Pregnant, lactating, or plans to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Study product-related Serious Adverse Events (SAEs) | 24 months
  Evaluate the safety of AMDC-GIR following treatment of tongue dysphagia
Study product-related, biopsy procedure-related, and injection procedure-related adverse events | 24 months
  Safety will be determined by the frequency and severity of adverse events related to study procedures and study product

SECONDARY OUTCOMES:
Penetration-Aspiration scale rating from swallowing fluoroscopy | 24 months
  Efficacy of AMDC-GIR in the improvement of objective fluoroscopic swallowing parameters
Pharyngeal Constriction Ratio measurement from swallowing fluoroscopy | 24 months
  Efficacy of AMDC-GIR in the improvement of objective fluoroscopic swallowing parameters
Upper Esophageal Sphincter opening measurement from swallowing fluoroscopy | 24 months
  Efficacy of AMDC-GIR in the improvement of objective fluoroscopic swallowing parameters
Pharyngeal transit time measurement from swallowing fluoroscopy | 24 months
  Efficacy of AMDC-GIR in the improvement of objective fluoroscopic swallowing parameters
Peak pharyngeal pressure measurement from high-resolution manometry | 24 months
  Efficacy of AMDC-GIR in the improvement of objective manometric swallowing parameters
Anterior tongue pressure measurement from Iowa Oral Performance Instrument (IOPI) | 24 months
  Efficacy of AMDC-GIR in the improvement of objective Anterior Tongue Pressure Measurement (IOPI)
Patient-reported dysphagia symptoms based on Eating Assessment Tool- EAT10 score | 24 months
  Effect of AMDC-GIR on patient-reported dysphagia symptoms [Eating Assessment Tool- EAT10]
Patient-reported quality of life based on SF-12 survey score | 24 months
  Effect of AMDC-GIR on patient-reported dysphagia symptoms quality of life (QOL) [SF-12]
Patient-reported voice symptoms based on Voice Handicap Index - VHI10 score | 24 months
  Effect of AMDC-GIR on patient-reported dysphagia symptoms and voice symptoms [Voice Handicap Index - VHI10]

CONTACTS AND LOCATIONS:
Overall Officials: Peter Belafsky, MD, PhD, Principal Investigator — University of California Davis, Department of Otolaryngology; Maggie Kuhn, MD, Principal Investigator — University of California Davis, Department of Otolaryngology; Nogah Nativ, PhD, Study Director — University of California Davis, Department of Otolaryngology
Locations (1):
- UC Davis Medical Center, Department of Otolaryngology, Head and Neck Surgery, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No